CLINICAL TRIAL: NCT01425073
Title: Discontinuation of Trimethoprim-sulfamethoxazole Prophylaxis in Adults on Antiretroviral Therapy in Kenya: a Randomized Trial
Brief Title: Discontinuation of Trimethoprim-sulfamethoxazole Prophylaxis in Adults on Antiretroviral Therapy in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Christina Polyak, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40461-B
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome; Disease Progression; Immune System Diseases; Malaria; Parasitic Diseases; Pneumonia; Diarrhea; Infectious Disorder of Immune System
Keywords: HIV; Co-Infections; Malaria; Pneumonia; Diarrhea
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Disease Progression; Immune System Diseases; Malaria; Parasitic Diseases; Pneumonia; Diarrhea; Coinfection | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stop TMP/SMZ (Experimental): Arm 1 will have patients discontinue trimethoprim-sulfamethoxazole (TMP/SMZ) prophylaxis; patients will follow up every 3 months with study staff.
  Interventions: Other: Discontinue TMP/SMZ prophylaxis
- Standard of care TMP/SMZ prophylaxis (No Intervention): Arm 2 will continue standard of care treatment with trimethoprim-sulfamethoxazole (TMP/SMZ) prophylaxis.

INTERVENTIONS:
Other: Discontinue TMP/SMZ prophylaxis — Subjects in the intervention arm will discontinue use of daily TMP/SMZ for the duration of the study
  Other Names: Septrin; Septra; Cotrimoxazole; Bactrim
  Arms: Stop TMP/SMZ

SUMMARY:
Both antiretroviral therapy (ART) and prevention of opportunistic infections (OIs) have been associated with significantly decreased mortality in HIV-infected individuals. Trimethoprim-sulfamethoxazole (TMP/SMZ), also known as bactrim, is a common antibiotic and used as prophylaxis for OIs. For countries with high prevalence of HIV and limited health infrastructure, the WHO endorses universal TMP/SMZ for all HIV-infected individuals. Notably, these guidelines were created prior to the scale-up of ARTs. Following ART and subsequent immune recovery, TMP/SMZ may no longer be required. In the US and Europe, for example, TMP/SMZ is discontinued after patients show evidence of immune recovery. Therefore, we propose a prospective randomized trial among HIV infected individuals on ART with evidence of immune recovery (ART for > 18mo and CD4 >350 cells/mm3) to determine whether continued TMP/SMZ prophylaxis confers benefits in decreasing morbidity (malaria, pneumonia, diarrhea), mortality, CD4 count maintenance, ART treatment failure and malaria immune responses.

DETAILED DESCRIPTION:
Please see summary above.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age.
* Participants must be willing to participate and give written informed consent.
* Participants must be willing and able to return for the scheduled follow-up visits.
* Participants must have been on ART for > 18 months.
* Participants must have a CD4 count of > 350 cells/mm3.
* Participants must not be suspected of ART treatment failure.

Exclusion Criteria:

* Participants must not be pregnant at enrollment (by urine HCG testing).
* Participants must not be breastfeeding at the time of enrollment.
* Participants must be on first-line ART therapy as defined by Kenyan National Guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incidence of severe infectious morbidity (malaria, pneumonia, diarrhea) | 12 months
  A combined outcome of malaria, pneumonia or severe diarrhea.

SECONDARY OUTCOMES:
CD4 count increase | 12 months
  CD4 count increase
Rate of ART treatment failure | 12 months
  Rate of ART treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Christina Polyak, MD, MPH, Principal Investigator — Kenya Medical Research Institute/ Department of Medicine, University of Washington
Locations (2):
- Kenya (2):
  - Homa Bay District Hospital, Homa Bay, Nyanza Pronvince
  - Kombewa District Hospital, Kombewa, Nyanza

REFERENCES:
- [Background] McNaghten AD, Hanson DL, Jones JL, Dworkin MS, Ward JW. Effects of antiretroviral therapy and opportunistic illness primary chemoprophylaxis on survival after AIDS diagnosis. Adult/Adolescent Spectrum of Disease Group. AIDS. 1999 Sep 10;13(13):1687-95. doi: 10.1097/00002030-199909100-00012. PMID 10509570
- [Background] Anglaret X, Chene G, Attia A, Toure S, Lafont S, Combe P, Manlan K, N'Dri-Yoman T, Salamon R. Early chemoprophylaxis with trimethoprim-sulphamethoxazole for HIV-1-infected adults in Abidjan, Cote d'Ivoire: a randomised trial. Cotrimo-CI Study Group. Lancet. 1999 May 1;353(9163):1463-8. doi: 10.1016/s0140-6736(98)07399-1. PMID 10232311
- [Background] Wiktor SZ, Sassan-Morokro M, Grant AD, Abouya L, Karon JM, Maurice C, Djomand G, Ackah A, Domoua K, Kadio A, Yapi A, Combe P, Tossou O, Roels TH, Lackritz EM, Coulibaly D, De Cock KM, Coulibaly IM, Greenberg AE. Efficacy of trimethoprim-sulphamethoxazole prophylaxis to decrease morbidity and mortality in HIV-1-infected patients with tuberculosis in Abidjan, Cote d'Ivoire: a randomised controlled trial. Lancet. 1999 May 1;353(9163):1469-75. doi: 10.1016/s0140-6736(99)03465-0. PMID 10232312
- [Background] Mermin J, Lule J, Ekwaru JP, Malamba S, Downing R, Ransom R, Kaharuza F, Culver D, Kizito F, Bunnell R, Kigozi A, Nakanjako D, Wafula W, Quick R. Effect of co-trimoxazole prophylaxis on morbidity, mortality, CD4-cell count, and viral load in HIV infection in rural Uganda. Lancet. 2004 Oct 16-22;364(9443):1428-34. doi: 10.1016/S0140-6736(04)17225-5. PMID 15488218
- [Background] Hamel MJ, Greene C, Chiller T, Ouma P, Polyak C, Otieno K, Williamson J, Shi YP, Feikin DR, Marston B, Brooks JT, Poe A, Zhou Z, Ochieng B, Mintz E, Slutsker L. Does cotrimoxazole prophylaxis for the prevention of HIV-associated opportunistic infections select for resistant pathogens in Kenyan adults? Am J Trop Med Hyg. 2008 Sep;79(3):320-30. PMID 18784222
- [Background] Furrer H, Egger M, Opravil M, Bernasconi E, Hirschel B, Battegay M, Telenti A, Vernazza PL, Rickenbach M, Flepp M, Malinverni R. Discontinuation of primary prophylaxis against Pneumocystis carinii pneumonia in HIV-1-infected adults treated with combination antiretroviral therapy. Swiss HIV Cohort Study. N Engl J Med. 1999 Apr 29;340(17):1301-6. doi: 10.1056/NEJM199904293401701. PMID 10219064
- [Background] Weverling GJ, Mocroft A, Ledergerber B, Kirk O, Gonzales-Lahoz J, d'Arminio Monforte A, Proenca R, Phillips AN, Lundgren JD, Reiss P. Discontinuation of Pneumocystis carinii pneumonia prophylaxis after start of highly active antiretroviral therapy in HIV-1 infection. EuroSIDA Study Group. Lancet. 1999 Apr 17;353(9161):1293-8. doi: 10.1016/s0140-6736(99)03287-0. PMID 10218526
- [Background] Lowrance D, Makombe S, Harries A, Yu J, Aberle-Grasse J, Eiger O, Shiraishi R, Marston B, Ellerbrock T, Libamba E. Lower early mortality rates among patients receiving antiretroviral treatment at clinics offering cotrimoxazole prophylaxis in Malawi. J Acquir Immune Defic Syndr. 2007 Sep 1;46(1):56-61. PMID 17972365
- [Background] Walker AS, Ford D, Gilks CF, Munderi P, Ssali F, Reid A, Katabira E, Grosskurth H, Mugyenyi P, Hakim J, Darbyshire JH, Gibb DM, Babiker AG. Daily co-trimoxazole prophylaxis in severely immunosuppressed HIV-infected adults in Africa started on combination antiretroviral therapy: an observational analysis of the DART cohort. Lancet. 2010 Apr 10;375(9722):1278-86. doi: 10.1016/S0140-6736(10)60057-8. Epub 2010 Mar 27. PMID 20347483
- [Background] Phillips-Howard PA, Nahlen BL, Kolczak MS, Hightower AW, ter Kuile FO, Alaii JA, Gimnig JE, Arudo J, Vulule JM, Odhacha A, Kachur SP, Schoute E, Rosen DH, Sexton JD, Oloo AJ, Hawley WA. Efficacy of permethrin-treated bed nets in the prevention of mortality in young children in an area of high perennial malaria transmission in western Kenya. Am J Trop Med Hyg. 2003 Apr;68(4 Suppl):23-9. PMID 12749482
- [Background] Piaggio G, Elbourne DR, Altman DG, Pocock SJ, Evans SJ; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: an extension of the CONSORT statement. JAMA. 2006 Mar 8;295(10):1152-60. doi: 10.1001/jama.295.10.1152. PMID 16522836
- [Derived] Juma DW, Muiruri P, Yuhas K, John-Stewart G, Ottichilo R, Waitumbi J, Singa B, Polyak C, Kamau E. The prevalence and antifolate drug resistance profiles of Plasmodium falciparum in study participants randomized to discontinue or continue cotrimoxazole prophylaxis. PLoS Negl Trop Dis. 2019 Mar 21;13(3):e0007223. doi: 10.1371/journal.pntd.0007223. eCollection 2019 Mar. PMID 30897090
- [Derived] Ottichilo RK, Polyak CS, Guyah B, Singa B, Nyataya J, Yuhas K, John-Stewart G, Waitumbi JN. Malaria Parasitemia and Parasite Density in Antiretroviral-Treated HIV-Infected Adults Following Discontinuation of Cotrimoxazole Prophylaxis. J Infect Dis. 2017 Jan 1;215(1):88-94. doi: 10.1093/infdis/jiw495. Epub 2016 Oct 25. PMID 28077587
- [Derived] Polyak CS, Yuhas K, Singa B, Khaemba M, Walson J, Richardson BA, John-Stewart G. Cotrimoxazole Prophylaxis Discontinuation among Antiretroviral-Treated HIV-1-Infected Adults in Kenya: A Randomized Non-inferiority Trial. PLoS Med. 2016 Jan 5;13(1):e1001934. doi: 10.1371/journal.pmed.1001934. eCollection 2016 Jan. PMID 26731191